CLINICAL TRIAL: NCT04203550
Title: The Finnish Study of Intraoperative Irrigation Versus Drain Alone After Evacuation of Chronic Subdural Hematoma (FINISH): a Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: The Finnish Study of Intraoperative Irrigation Versus Drain Alone After Evacuation of Chronic Subdural Hematoma (FINISH)
Acronym: FINISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Kimmo Lonnrot, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3035/2019
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural hematoma; Surgical evacuation; Recurrence; Irrigation fluid
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, parallel group non-inferiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the treatment, it is not possible to blind the surgeon and OR staff from the treatment allocation. Measures to minimize bias include:
  * The patient will not be informed of treatment allocation
  * Treatment allocation will not be documented in medical records i.e. all the personnel participating in patient care after operation will be blinded to allocation
  * The study group members collecting postoperative data and performing the statistical analyses will be blinded to treatment arm until the analyses are finished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigation group (IR) (Active Comparator): A burr-hole craniostomy is performed and the dura is opened sharply and 10 ml of subdural exudate is aspired with blunt aspiration needle for a CSDH sample to be stored in -70℃ to be used for later analysis. Subdural space is irrigated by repeated rinsing with body temperature saline solution with a syringe and blunt needle until surgeon considers exudate to be clear. Minimum volume of irrigation will be 200 ml per operated side. The subdural drain is inserted 3-5 cm underneath the skull and parallel to it. The total volume of irrigation as well as the duration of operation is recorded.
  Interventions: Procedure: Intraoperative irrigation
- No-Irrigation group (N-IR) (Experimental): A burr-hole craniostomy is performed and a small incision to the dura is made and 10 ml of subdural exudate is aspired with blunt aspiration needle for a CSDH sample to be stored in -70℃ to be used for later analysis. The subdural drain is inserted approximately 3-5 cm underneath the skull and parallel to it. The duration of operation is recorded.
  Interventions: Procedure: No irrigation

INTERVENTIONS:
Procedure: Intraoperative irrigation — Operation with irrigation
  Arms: Irrigation group (IR)
Procedure: No irrigation — Operation without irrigation
  Arms: No-Irrigation group (N-IR)

SUMMARY:
FINISH-trial is a prospective, randomized, controlled, parallel group non-inferiority trial comparing single burr-hole evacuation of chronic subdural hematoma (CSDH) with intraoperative irrigation (IR) and evacuation of CSDH without irrigation (N-IR).

DETAILED DESCRIPTION:
FINISH-trial is a prospective, randomized, controlled, parallel group non-inferiority trial comparing single burr-hole evacuation of chronic subdural hematoma (CSDH) with intraoperative irrigation (IR) and evacuation of CSDH without irrigation (N-IR). In both groups, a passive subdural drain is used for 48 hours as a standard of treatment. The study will be conducted in all five neurosurgical departments in Finland. To determine whether operation without irrigation results in non-inferior outcome to operation with irrigation, we will randomize 426 patients into two groups and follow them up for 6 months using recurrence rates as the primary outcome. Secondary outcomes in our study include mortality, neurological outcome and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic unilateral or bilateral CSDH requiring burr-hole evacuation

  o Predominantly hypodense or isodense on imaging (CT/MRI).
* Clinical symptoms correlating with the CSDH
* Patients with bilaterally operated CSDHs will be treated with the same protocol on both sides and analyzed as a single study participant

Exclusion Criteria:

* CSDH requiring surgical treatment other that burr-hole evacuation (e.g. craniotomy)
* CSDH in a patient who has a cerebrospinal fluid shunt
* Patients who have undergone any intracranial surgery before
* Comatose patients (GCS 8 or lower) with absent motor responses to painful stimuli; decerebrate or decorticate posturing
* Patient's postoperative cooperation is suspected to be insufficient for drain usage, i.e. disoriented or semiconscious patient
* Patient has a hematogenic malignancy that has obtained active treatment within the previous five years
* Patient has a central nervous system tumor or malignancy
* Patient has acute infection with fever and requires antibiotic treatment at the moment
* Patient has a high risk of life-threatening thrombosis (e.g. recent coronary stent, recent pulmonary embolism, low cardiac valve replacement) and discontinuation of antithrombotic medication is not recommended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Rate of re-operations of ipsilateral chronic subdural hematoma | From operation up to 6 months after postoperatively
  Rate of reoperations between groups

SECONDARY OUTCOMES:
Change of Modified Rankin Scale (MRS) from baseline to 6 months after operation | At baseline, and at 2 and 6 months after operation
  Modified Rankin scale ranges from 1 to 6, where 1 indicates normal daily functionality and 6 indicates death
Rate of mortality between intervention groups | From operation up to 6 months postoperatively
  Rate of mortality between intervention groups
Duration of the operation between groups | Intraoperative measure
  Time (minutes) used to complete the operation, from incision to last suture
Hospital length of stay between groups | From operation up to six months
  The duration of the stay in hospital (days)
Change in the volume of CSDH in the CT or MRI image between baseline and 2 months post-operatively | Immediate preoperative and 2 months postoperatively
  The volume of CSDH will be measured from preoperative CT or MRI and at 2 months after operation CT or MRI
Rate of complications and adverse events within 6 months | within 6 months after operation
  Rate of complication rate between groups

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Lönnrot, MD, Ph.D, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) is available upon request when General Data Protection Regulation (GDPR) and guiding legislation regulations are fulfilled.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol and Statistical Analysis Plan (SAP) will be published after the study has started. Other document will be available as study proceeds and after study is completed.
Access Criteria: Data access request will be reviewed by FINISH-trial steering group. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Tommiska P, Knuutinen O, Lonnrot K, Luoto T, Leinonen V, Koivisto T, Tetri S, Posti JP, Raj R; FINISH study group. Mortality and causes of death after surgery for chronic subdural hematoma: a post hoc study of the FINISH randomized trial. Acta Neurochir (Wien). 2025 Dec 1;167(1):310. doi: 10.1007/s00701-025-06728-9. PMID 41326886
- [Derived] Knuutinen O, Maatta J, Kovalainen A, Pohjola A, Tommiska P, Raj R; FINISH study group. Surgical Delay and Functional Outcome After Surgery for Chronic Subdural Hematoma. World Neurosurg. 2025 May;197:123843. doi: 10.1016/j.wneu.2025.123843. Epub 2025 Feb 28. PMID 40024327
- [Derived] Tommiska P, Knuutinen O, Lonnrot K, Kivisaari R, Raj R; FINISH study group. Association between postoperative thromboembolic and hemorrhagic complications and clinical outcomes after surgery for chronic subdural hematoma in patients with anticoagulation therapy for atrial fibrillation. Acta Neurochir (Wien). 2025 Jan 16;167(1):17. doi: 10.1007/s00701-024-06417-z. PMID 39815109
- [Derived] Raj R, Tommiska P, Koivisto T, Leinonen V, Danner N, Posti JP, Laukka D, Luoto T, Rauhala M, Tetri S, Korhonen TK, Satopaa J, Kivisaari R, Luostarinen T, Schwartz C, Czuba T, Taimela S, Lonnrot K, Jarvinen TLN; Finnish study of intraoperative irrigation versus drain alone after evacuation of CSDH (FINISH) study group. Burr-hole drainage with or without irrigation for chronic subdural haematoma (FINISH): a Finnish, nationwide, parallel-group, multicentre, randomised, controlled, non-inferiority trial. Lancet. 2024 Jun 29;403(10446):2798-2806. doi: 10.1016/S0140-6736(24)00686-X. Epub 2024 Jun 6. PMID 38852600
- [Derived] Tommiska P, Raj R, Schwartz C, Kivisaari R, Luostarinen T, Satopaa J, Taimela S, Jarvinen T, Ranstam J, Frantzen J, Posti J, Luoto TM, Leinonen V, Tetri S, Koivisto T, Lonnrot K. Finnish study of intraoperative irrigation versus drain alone after evacuation of chronic subdural haematoma (FINISH): a study protocol for a multicentre randomised controlled trial. BMJ Open. 2020 Jun 21;10(6):e038275. doi: 10.1136/bmjopen-2020-038275. PMID 32565480

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT04203550/SAP_000.pdf